CLINICAL TRIAL: NCT06825936
Title: Asian-Mediterranean Diet and Women's Health: A Randomized Controlled Trial (A+ MEAL Study)
Brief Title: Asian-Mediterranean Diet and Women's Health
Acronym: A+ MEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Global Centre for Asian Women's Health (Other)
Collaborators: Yong Loo Lin School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-371
Record Dates: First submitted 2025-02-06; First posted 2025-02-13 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cardiometabolic Risk Factors; Cardiometabolic Conditions; Women Health
Keywords: Cardiometabolic health; Mediterranean diet; Women health; Cardiometabolic risk factors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Diet intervention consisting of study meals and nuts along with diet advice
  Interventions: Other: Diet intervention
- Control (Placebo Comparator): Diet advice following national guidelines
  Interventions: Other: Control

INTERVENTIONS:
Other: Diet intervention — For participants assigned to the intervention arm, the dietary intervention consists of: a) pre-cooked Asian-Mediterranean meals: participants will receive free meals, two meals a day, five days a week, and b) pre-packed nuts, 30g a day, five days a week, during the intervention period. Additionally, participants will receive a dietary consultation session at baseline and every four weeks.
  Arms: Intervention
Other: Control — For participants assigned to the control arm, they will receive a leaflet with dietary advice based on national guidelines at baseline.
  Arms: Control

SUMMARY:
Given the escalating high burdens of overeight and obesity, and related commobidies in Asia, Asian women with overweight/obesity is an important group for targeted intervention in promoting health and wellbeing. A study focused on Asian women at reproductive or early post-menopausal age can inform effective strategies for promoting healthy diet and lifetyle and for optimizing health not only among these women but also for their children and partners.

The Mediterranean diet has beneficial effects on cardiometabolic and reproductive health. So far, evidence on the Mediterranean diet and its health benefits mostly come from Western populations. Studies evaluating health effects of Mediterranean diet in Asian population are scant.

This study aims to investigate the beneficial effects of a healthy, Mediterranean-inspired localized diet (i.e., Asian-Mediterranean diet) on women's health, such as cardiometabolic health with potential mechanisms through modulating gut and brain health.

DETAILED DESCRIPTION:
This study is a two-arm, single-centre, randomized controlled trial (RCT) involving up to 300 women of Chinese ethnicity in Singapore between 21-50 years old. Upon enrollment, participants will be randomized into one of two study arms (Intervention (up to 150 women), Control (up to 150 women)) in 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the inclusion criteria for participation:

1. Females aged 21-50 years
2. Chinese ethnicity
3. Singapore citizens, permanent residents, or long-term pass holders
4. Is able to complete questionnaires in English
5. BMI ≥ 23.0 kg/m2 but < 37.5 kg/m2
6. Not planning to conceive in the next 12 months from enrolment (you will be asked to withdraw once you conceive during the study period)
7. Not planning to leave Singapore for more than 2 consecutive calendar weeks (10 working days) in the next six months from enrolment
8. Not currently pregnant or breastfeeding
9. Not currently smoking
10. Without history of major chronic diseases (e.g., cancer, diabetes, cardiovascular diseases, chronic kidney disease), major infectious diseases (e.g. hepatitis B, HIV), severe gastrointestinal disorders (e.g. colitis or inflammation of the bowel, celiac disease, chronic gastritis) and major medical procedures/surgeries related to these conditions
11. Without major mental health condition
12. Without known food allergies, especially to nuts and seafood.
13. Not on any special diets or having dietary restrictions (e.g. vegetarians, vegans, ketogenic, Kosher diet)
14. Not currently and will not be enrolled in another interventional study or studies that may affect weight, cardiometabolic health, gut, or brain health in the next six months from enrolment

Exclusion Criteria:

Subjects not meeting any of the above inclusion criteria will be excluded from participation.

Additional Exclusion Criteria for MRI procedure only:

i. Shoulder width ≥60cm ii. Has any medical implants or foreign bodies, particularly related to heart, brain, or eye implants, including but not limited to pacemakers, artificial heart valves, implantable cardioverter defibrillators, ventricular assist devices, brain stimulation devices, intrauterine devices, and breast biopsies (if any implant or tissue marker has been placed) iii. History of head injury or trauma with loss of consciousness iv. Metallic dental braces or dental implants v. Having claustrophobia vi. Drinks more than 30 units of alcohol per week (1 unit = 25mL 40% spirit, 1 can of beer = 2 units, 1 standard glass of wine = 2 units)

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
High-density lipoprotein cholesterol (HDL-C) | week 0, week 12, and up to week 20
  High-density lipoprotein cholesterol (HDL-C) in mg/dL (blood draw)
Low-density lipoprotein cholesterol (LDL-C) | week 0, week 12, and up to week 20
  Low-density lipoprotein cholesterol (LDL-C) in mg/dL (blood draw)
Low-density lipoprotein cholesterol (LDL-C) to high-density lipoprotein cholesterol (HDL-C) ratio | week 0, week 12, and up to week 20
  Low-density lipoprotein cholesterol (LDL-C) in mg/dL and high-density lipoprotein cholesterol (HDL-C) in mg/dL (blood draw) to derive LDL-C to HDL-C ratio
Triglycerides | week 0, week 12, and up to week 20
  Triglycerides in mg/dL (blood draw)
Interleukin-6 (IL-6) | week 0, week 12, and up to week 20
  Interleukin-6 (IL-6) in pg/mL (blood draw)
C-reactive protein (CRP) | week 0, week 12, and up to week 20
  C-reactive protein (CRP) in mg/L (blood draw)

CONTACTS AND LOCATIONS:
Overall Officials: Cuilin Zhang, MD, MPH, PhD, Principal Investigator — Global Centre for Asian Women's Health, Yong Loo Lin School of Medicine, National University of Singapore
Locations (1):
- Global Centre for Asian Women's Health, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
We will make a decision on IPD sharing as our trial further progresses.